CLINICAL TRIAL: NCT07082894
Title: The Effect of Preoperative Oral Magnesium on Emergence Agitation in Children Undergoing Adenotonsillectomy: A Double Blind Randomized Placebo Controlled Study
Brief Title: Effect of Preoperative Oral Magnesium on Emergence Agitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Radwa Emad Eissa, lecturer of anesthesiology, surgical intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR1217/5/25
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Magnesium; Emergence Agitation; Adenotonsillectomy
MeSH Terms: conditions — Emergence Delirium | interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium group (Experimental): cases will receive preoperative oral magnesium dose of 120 mg at one hour before surgery
  Interventions: Drug: Magnesium
- Control group (Placebo Comparator): cases will receive oral lemon juice at one hour before surgery.
  Interventions: Other: Placebo control

INTERVENTIONS:
Drug: Magnesium — preoperative oral magnesium dose of 120 mg at one hour before surgery will be given.
  Arms: Magnesium group
Other: Placebo control — preoperative oral lemon juice at one hour before surgery will be given.
  Arms: Control group

SUMMARY:
This prospective randomized controlled study will be conducted to evaluate the effects of preoperative oral magnesium on the incidence and severity of emergence agitation in children undergoing adenotonsillectomy using sevoflurane anesthesia.

DETAILED DESCRIPTION:
Emergence agitation is a frequent postoperative complication in pediatric patients receiving inhalational anesthetics with a rapid recovery profile, e.g. sevoflurane. There is a wide variation in the reported incidence, with estimates ranging from 30% to 80%, depending on the definition, assessment tool and time frame of monitoring in the recovery period. Magnesium is a non-anesthetic N-methyl-D-aspartate receptor antagonist, which is as an anesthetic- and analgesic-sparing medication, with controversial clinical effectiveness. Regarding its use as a preventive measure against emergence agitation in children, only intraoperative intravenous route was studied and the results of previous reports were inconsistent. Oral magnesium syrup is a common drug used for enzyme activation, muscle and bone health, with calming effect and central nervous system supporting value.

In this novel study, the investigators will use magnesium via oral route before surgery as they hypothesize that the pre-emptive administration of the drug may decrease emergence agitation incidence in children undergoing adenotonsillectomy. Given the fact that preoperative anxiety and parent separation are predictors for emergence agitation, the calming effect, sleep promoting value of oral magnesium that may be obtained before anesthetic induction together with its peri-operative analgesic effects may explain its prophylactic benefit against emergence agitation.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* 4 to 7 years age
* American Society of Anesthesiologists (ASA) Physical Status I or II
* Scheduled for adenotonsillectomy surgery under sevoflurane anesthesia

Exclusion Criteria:

* Parents declined to participate in the trial
* Children with behavioral changes; neurological or psychiatric diseases
* Physical or developmental delay
* Sedative or anticonvulsant medication
* Pre-existing renal or cardiovascular disease, bone disease, or gastrointestinal disorders
* Allergy to magnesium

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence agitation | Up to 1 hour after surgery.
  Pediatric Anesthesia Emergence Delirium scale scores will be used and a score ≥ 10 will be considered to be a diagnostic endpoint for the development of agitation. It will be assessed on arrival to the post anesthesia care unit (PACU), and every 15 min thereafter for 1 hour

SECONDARY OUTCOMES:
Parental separation anxiety | Perioperative
  It will be assessed at the time of taking the child to the operating theater by the attending anesthesiologist using the Parent Separation Anxiety Scale. It ranges from one to four where one refers to easy separation; two equals whimpers; three denotes that the child cries and cannot be easily reassured, but not clinging to parents; and 4 signifies crying and clinging to parents. A score of 1 or 2 will be considered as 'acceptable' separation
Mask Acceptance Score | Perioperative
  Ease of mask acceptance will be graded using the Mask Acceptance Score. It is a 4-point scale: 1 = excellent (unafraid, accepts mask readily); 2 = good (slight fear of mask, easily reassured); 3 = fair (moderate fear of mask, not calmed with reassurance); and 4 = poor (terrified, combative and crying). A score of 1 or 2 will be considered 'satisfactory' mask acceptance
Postoperative pain | Up to 1 hour after surgery.
  the Face, Legs, Activity, Cry and Consolability (FLACC) scale will assess the pain degree at PACU arrival and every 0.25 hour for 1 hour after surgery. A FLACC score of at least 4 will be treated with 0.5mcg/kg of IV fentanyl.
Total dose of rescue fentanyl | Up to 1 hour after surgery.
  Fentanyl will be given for agitation or pain
Pediatric Anesthesia Emergence Delirium scale scores | Up to 1 hour after surgery.
  severity of agitation will be assessed by Pediatric Anesthesia Emergence Delirium scale.
Number of patients who will develop postoperative nausea and vomiting. | Up to 2 hours after surgery.
  Any episodes of nausea and vomiting will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available upon a reasonable request from the corresponding author after the end of the study for 1 year
Access Criteria: The data will be available upon a reasonable request from the corresponding author